CLINICAL TRIAL: NCT06415721
Title: Developing Functional Connectivity-Guided TMS for Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Collaborators: Stanford University (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Daniel McCalley, Postdoctoral Fellow, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PADNEW_0003
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse; Alcoholism; Drinking Behavior; Drinking Problem
Keywords: Transcranial Magnetic Stimulation; Veterans; Neuroimaging; Relapse
MeSH Terms: conditions — Alcoholism; Drinking Behavior; Recurrence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active fMRI-guided TMS (Experimental)
  Interventions: Device: Active Transcranial Magnetic Simulation
- Sham fMRI-guided TMS (Sham Comparator)
  Interventions: Device: Sham

INTERVENTIONS:
Device: Active Transcranial Magnetic Simulation — 1 session of active continuous theta burst stimulation (3600 pulses, 110% RMT) will be delivered to the cortical region demonstrating maximal functional connectivity with the striatum during alcohol cue presentation. TMS will be delivered using the Magventure MagPro X100.
  Other Names: MagVenture MagPro X100; Continuous Theta Burst Stimulation
  Arms: Active fMRI-guided TMS
Device: Sham — 1 session of sham continuous theta burst stimulation (3600 pulses, 110% RMT) will be delivered to the cortical region demonstrating maximal functional connectivity with the striatum during alcohol cue presentation. The MagVenture MagPro x100 is capable of administering a sham stimulation. The reverse side of the TMS coil is plated with a magnetic shield such that electromagnetic energy cannot stimulate the brain. The device offers compatibility with Transcutaneous Electrical Nerve Stimulation devices such that titrated electrical pulses can be delivered to the scalp location to mimic the sensation of a TMS pulse without stimulating the brain.
  Other Names: MagVenture MagPro X100
  Arms: Sham fMRI-guided TMS

SUMMARY:
Alcohol Use Disorders are currently positioned as the third leading cause of preventable death in the United States, constituting a humanitarian crisis with substantial financial burden on society and medical facilities. While several pharmacological interventions exist, 60% of individuals who seek these treatments relapse to alcohol within 6 months. These high relapse rates are due in part to elevated brain response to alcohol cues in the environment. This study seeks to evaluate the efficacy of one session of functional Magnetic Resonance Imaging (fMRI) guided transcranial magnetic stimulation (TMS) as a strategy to reduce brain reactivity to alcohol cues.

DETAILED DESCRIPTION:
At least 60% of those with AUD will experience a major relapse period within 6 months of treatment, irrespective of the intervention (psychosocial and/or pharmacological) employed. Consequently, the high prevalence of AUD and relapse following treatment in Veterans is associated with substantial resource allocation and costs for the VA Health Care System. Current pharmacological and psychosocial interventions demonstrate only a moderate level of efficacy, which is reflected in the high rate of relapse in AUD. Transcanial Magnetic Stimulation (TMS) is a neurostimulation method that is at the forefront of innovative, non-invasive, and safe treatments for AUD, and other psychiatric disorders. To reduce the high rate of relapse in Veterans with AUD, it is necessary for interventions to more effectively address the associated neurobiological dysfunction. Non-invasive neuromodulation techniques are showing promise toward the aim of modifying specific and selective neural targets related to AUD and relapse. To date, TMS has been primarily delivered to the dorsolateral and medial prefrontal cortices as these regions are, on average, highly reactive to alcohol cues. On an individual basis, however, peak brain response to alcohol cues can vary substantially in spatial location within the brain. Retrospective analyses of TMS-AUD clinical trails has demonstrated that when TMS is delivered to an individual's peak brain response to alcohol cues, the likelihood of remaining abstinent is increased by a factor of 5.6 (relative to sham TMS treatment). This study aims to deliver one session of TMS to a cortical target which displays peak functional connectivity to the ventral striatum, a key brain region mediating reward and alcohol cue reactivity. The ultimate goal of this study evaluate change in brain reactivity to alcohol cues following active and sham TMS.

ELIGIBILITY:
Inclusion Criteria:

* Between age 25 and 75.
* Current DSM-5 diagnosis of moderate to severe AUD (≥4 diagnostic symptoms).
* Able to attend scheduled clinic visits
* Able to read, understand and voluntarily sign Informed Consent prior to participating in any study-specific procedures or assessments.
* If on a medication regimen, that regimen will be stable for the duration of the study;
* Fluency in English.

Exclusion Criteria:

* Transcranial magnetic stimulation (TMS) and magnetic resonance imaging (MRI) contraindications: such as a cardiac pacemaker, cochlear implant, or an implanted device (deep brain stimulation, metal in the head, metal in the body, claustrophobia, pregnant or breastfeeding or other ferromagnetic device/objected in the head and body within 30 cm of the treatment coil.
* General medical condition, disease or neurological disorder that interferes with the assessments or participation.
* Unable to safely withdraw, at least two weeks prior to treatment, from medications that increase seizure risk.
* Current substance abuse (except caffeine or nicotine) as determined by positive toxicology screen.
* Have a mass lesion, cerebral infarct, or other active CNS disease, including an alcohol-related seizure or a seizure disorder. • A recent suicide attempt (defined as within the last 30 days) or presence of current suicidal plan or intent. Patients at risk for suicide will be required to establish a written safety plan involving their primary therapist before entering the study.
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to follow study protocols. • Greater than mild traumatic brain injury (defined as greater than 10 minutes loss of consciousness).
* Taking benzodiazepine or neuroleptic medications, or any medication known to alter seizure threshold
* unstable chronic illness.
* Current or lifetime history of bipolar disorder or psychosis.
* Participation in another concurrent intervention based clinical trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in blood-oxygen level dependent signal as a measure of change in alcohol cue reactivity | Baseline (pre-TMS) and Day 2 (post-TMS)
  The effect of real versus sham fMRI-guided TMS on alcohol cue reactivity will be assessed by comparing brain reactivity to images of alcohol ('alcohol cues') shown during the fMRI scan. Change in blood-oxygen level dependent signal magnitude will be measured within the striatum, a key brain region involved in cue-reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McCalley, PhD, Principal Investigator — Palo Alto VA Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data, specimens, forms, reports and other records that leave the site will be identified only by a participant ID number to maintain confidentiality. The ID Number will have no relationship to any aspect of identifiable private information. Therefore, the data associated with each participant will be completely de-identified and there will be no mechanism by which users can re-identify participant data with the subject code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three to twelve months after publication
Access Criteria: Researchers who provide a methodologically sound proposal.